CLINICAL TRIAL: NCT05926297
Title: Treatment of Peri-implant Mucositis by Non-surgical Debridement and Adjunctive Application of a Combination of Sodium Hypochlorite Gel and Cross-linked Hyaluronic Acid Gel
Brief Title: Treatment of Peri-implant Mucositis by Sodium Hypochlorite Gel and Cross-linked Hyaluronic Acid Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Clinical Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110/2023; 140/2023 (Other: Semmelweis University, Faculty of Dentistry)
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-03

CONDITIONS: Peri-implant Mucositis; Mucositis Oral
Keywords: Hyaluronic Acid; Peri-implant mucositis; Sodium hypochlorite
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: The study will be designed as a double-arm randomized controlled clinical trial. Mucositis will be treated with NaOCl-based gel + NSMD + HA-based gel in Test group and with NSMD alone in Control group. All clinical parameters will be recorded and the final evaluation will be performed.
Who Masked: Participant
Masking Description: Only patients will be unaware of the type of treatment performed, with prior written informed consent. So, they will be divided in the two groups of study after a process of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NaOCl + HA Group (Experimental): A NaOCl-based gel will initially be applied in the peri-implant sulcus for 30 seconds, without the need for flushing. Furthermore, mechanical therapy (NSMD) will be performed by means of an ultrasonic scaler with a plastic tip. Finally, the HA-based gel will be applied in the peri-implant sulcus by means of a blunt-tipped needle.
  Interventions: Procedure: Application NaOCl gel + HA gel
- NSMD Group (Active Comparator): Control group will be treated only through a non-surgical mechanical therapy with curettes or scaler tips.
  Interventions: Procedure: Non-surgical mechanical debridement

INTERVENTIONS:
Procedure: Application NaOCl gel + HA gel — First step: application of NaOCl gel Second step: NSMD Third step: application of HA gel
  Arms: NaOCl + HA Group
Procedure: Non-surgical mechanical debridement — Only mechanical debridement with curettes ans scaler tips
  Arms: NSMD Group

SUMMARY:
The aim of the study is to evaluate the potential of the combination of a sodium hypochlorite-based gel and a hyaluronic acid-based gel as an adjuvant to Non-Surgical Mechanical Debridement (NSMD) in the treatment of mucositis, after 6 months of follow-up. After a meticulous selection, patients will be randomly assigned to Test (Sodium Hypochlorite-based gel + NSMD + Hyaluronic Acid-based gel ) or Control (NSMD) group. All clinical parameters will be recorded and the final evaluation will be performed.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the clinical results of the combination of a sodium hypochlorite-based gel (NaOCl gel) and a cross-linked hyaluronic acid-based gel (HA gel) as an adjuvant to Non-Surgical Mechanical Debridement (NSMD) in the treatment of mucositis, after 6 months of follow-up (Clean & Seal concept). Following the selection through inclusion and exclusion criteria, all patients will be randomly assigned to Test NaOCl-based gel + NSMD + HA-based gel) or Control (NSMD) group.

Patients will be recruited at Department of Periodontology (Univeristy of Naples "Federico II") and at Department of Periodontology (University of Budapest "Semmelweis").

Subsequently, after recording of the clinical parameters (BoP, FMPS, FMBS, PD), in the Test group a NaOCl-based gel will initially be applied in the peri-implant sulcus for 30 seconds, without the need for flushing. Furthermore, mechanical therapy (NSMD) will be performed by means of an ultrasonic scaler with a plastic tip. Finally, HA-based gel will be applied in the peri-implant sulcus by means of a blunt-tipped needle. Conversely, Control group will be treated only through the NSMD.

All clinical parameters (BoP, FMPS, FMBS, PD) will be recorded again after 6 months for the final evaluation. Data analysis will be performed using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Non-smokers and smokers ( ≤ 10 cigarettes/day);
* Presence of at least 1 implant in mucositis, clinically and radiographically detected;
* The implant in mucositis (tissue-level or bone-level) must support a fixed prosthetic device (single crown, 3-element bridge), cemented or screwed.

Exclusion Criteria:

* Cancer patients;
* Uncontrolled diabetic patients;
* Prolonged antibiotic treatment or anti-inflammatory treatment in the previous 6 months;
* Pregnant or breastfeeding patients;
* Implants that support mobile prosthetic products;
* Implants in peri-implantitis, detected clinically and radiographically.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change of BoP (+/-) | baseline, 6 months after periodontal therapy
  Bleeding on periodontal probing

SECONDARY OUTCOMES:
Change of Full-mouth Plaque Score (FMPS; %) | baseline, 6 months after periodontal therapy
  Percentage of all sites exhibiting plaque
Change of Full-mouth Bleeding Score (FMBS; %) | baseline, 6 months after periodontal therapy
  Percentage of all sites exhibiting bleeding
Change of Probing Depth (PD; millimeters). | baseline, 6 months after periodontal therapy
  Distance from the gingival margin to the bottom of the peri-implant pocket

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ramaglia, Principal Investigator — Federico II University
Locations (2):
- Semmelweis University, Budapest, HU, Hungary
- University of Naples Federico II, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: No